CLINICAL TRIAL: NCT00236808
Title: A Multicenter, Double-Blind Study to Compare the Safety and Efficacy of Levofloxacin to That of Ciprofloxacin in the Treatment of Chronic Prostatitis
Brief Title: A Study to Evaluate the Safety and Effectiveness of Levofloxacin Compared With Ciprofloxacin in Patients With Chronic Bacterial Prostatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005551
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Prostatitis
Keywords: quinolones, ciprofloxacin; levofloxacin; chronic bacterial prostatitis; inflammation; chronic prostatitis; prostatitis; prostate; antibiotic
MeSH Terms: conditions — Prostatitis; Inflammation | interventions — Levofloxacin

INTERVENTIONS:
Drug: levofloxacin

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of levofloxacin to ciprofloxacin in patients with chronic bacterial prostatitis.

DETAILED DESCRIPTION:
Prostatitis (an inflammation of the prostate) is the most common condition affecting the urinary system in men under 50 years of age. Symptoms of chronic (long-term) prostatitis may include urgency to urinate, frequency or difficulty in urinating or abdominal, pelvic, or rectal pain. A frequent cause of prostatitis is bacterial infection, treatable with antibiotics. This multicenter, double-blind study evaluates the safety and effectiveness of levofloxacin as compared to ciprofloxacin in patients with chronic bacterial prostatitis. Patients receive treatment with either levofloxacin or ciprofloxacin for 28 days and are evaluated during treatment and 5-12 days after the last dose of study drug (posttherapy visit), and 1 month after the last dose (poststudy visit). Patients are contacted six months after the last dose to follow up on the potential recurrence of their prostatitis. Effectiveness is assessed by measuring the ability of the study drug to eliminate bacteria causing prostatitis and to reduce the signs and symptoms of chronic prostatitis. Laboratory tests for presence of bacteria are performed throughout the study and at each visit, patients are questioned as to the relief of their symptoms. Safety evaluations (incidence of adverse events, physical examinations, laboratory tests) are performed throughout the study. The study hypothesis is that levofloxacin is at least as effective as ciprofloxacin in treating chronic bacterial prostatitis without any significant safety issues being observed.

Levofloxacin 500 milligrams (mg) by mouth once daily or ciprofloxacin 500 mg by mouth twice daily for 28 days

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic prostatitis meeting all 3 of the following criteria: 1) clinical signs and symptoms of prostatitis including tender prostate and one or more of the following: difficulty in, frequency of, or urgency of urinating, retention of urine or hesitancy in urinating, decreased urinary stream, painful ejaculation, pelvic or low back pain, pain on examination, fever or chills
* 2) history of chronic prostatitis defined as 1 previous episode lasting 4 weeks or 2 or more episodes during the previous 12 months
* And 3) laboratory evidence of prostatitis
* Able to take oral medications
* Over-the-counter medications for chronic prostatitis are continued at the same dose during the study or are discontinued before study entry

Exclusion Criteria:

* Have taken an antibiotic similar to levofloxacin for any reason within the past 14 days
* Have received any medication for more than 24 hours during the past 7 days that may be effective in treating prostatitis unless there is evidence of treatment failure after 5 or more days of treatment with the other medication
* Have had certain surgeries during the past 6 months, including prostate surgery, surgical opening of the bladder or kidney or insertion of a permanent catheter (tube) for urination
* Taking any medications that may affect bladder or prostate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2000-05; Study Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
Microbiologic eradication of bacteria at posttherapy visit

SECONDARY OUTCOMES:
Clinical response rates based upon signs and symptoms at posttherapy and poststudy; microbiologic eradication of bacteria at poststudy; Incidence of adverse events, changes in physical examinations, vital signs, laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Bundrick W, Heron SP, Ray P, Schiff WM, Tennenberg AM, Wiesinger BA, Wright PA, Wu SC, Zadeikis N, Kahn JB. Levofloxacin versus ciprofloxacin in the treatment of chronic bacterial prostatitis: a randomized double-blind multicenter study. Urology. 2003 Sep;62(3):537-41. doi: 10.1016/s0090-4295(03)00565-x. PMID 12946763
- See also: A study to evaluate the safety and effectiveness of levofloxacin compared with ciprofloxacin in patients with chronic bacterial prostatitis. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=662&filename=CR005551_CSR.pdf